CLINICAL TRIAL: NCT02333994
Title: Efficacy of Education With Balance Exercise in Improving Balance and Reducing the Fear of Falls in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, DIVYA MIDHA, ASSISTANT PROFESSOR, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3456
Record Dates: First submitted 2015-01-01; First posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Distorted; Balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GROUP A (Experimental): EDUCATION PROGRAMME AND BALANCE TRAINING EXERCISES
  Interventions: Device: GROUP A education programme as well as balance training exercises
- GROUP B (Active Comparator): BALANCE EXERCISES
  Interventions: Other: GROUP B on-platform training

INTERVENTIONS:
Device: GROUP A education programme as well as balance training exercises — Group A received education programme as well as balance training exercises.The intervention group attended one-hour training classes once a week for 6 consecutive weeks. The classes involved both lectures and discussions and were guided through with handouts and worksheets. Each session began by giving a summary of the previous session and continued with the main topic of the session. The intervention program also engaged the participants in discussions about their concerns regarding falling and on topics pertaining to identifying and reducing the risk factors of falls, including environmental hazards in and out of the house
  Arms: GROUP A
Other: GROUP B on-platform training — on-platform training was performed while standing and while sitting on a 22-inch therapeutic ball, 1 eyes open or closed 2 normal or reduced area of foot support 3 on foam or floor 4 with or without manual p
  Other Names: BALANCE TRAINING
  Arms: GROUP B

SUMMARY:
The aim of the study was to evaluate the Efficacy of Education With Balance Exercise in Reducing Fear of Falls in Elderly Population . In the present study the educational program along with balance training was delivered to group A, (Experimental group) and only Balance training was delivered to group B, (Control group) for 6 weeks for 1 hr duration once weekly. Education program included education about the risk factors of falls such as environmental hazards, importance of good nutrition, use of stick while walking, avoiding slippery surfaces. Balance training consists of stance activities and balance exercise program. The outcome measures for this intervention were Activities specific balance confidence scale and berg balance scale.

DETAILED DESCRIPTION:
Present study was an experimental design. A total of 60 elderly subjects were selected as per the selection criteria and they were randomly allocated in two equal groups i.e.Group A- (Experimental Group)- Balance Exercises and Education Program Group B - (Control Group) - Balance exercises.procedure of study was explained to each subject and written consent was taken from them.

Aim:

The aim of the study was to evaluate the Efficacy of Education With Balance Exercise in Reducing Fear of Falls in Elderly Population .

Materials and Methods In the present study the educational program along with balance training was delivered to group A, (Experimental group) and only Balance training was delivered to group B, (Control group) for 6 weeks for 1 hr duration once weekly. Education program included education about the risk factors of falls such as environmental hazards, importance of good nutrition, use of stick while walking, avoiding slippery surfaces. Balance training consists of stance activities and balance exercise program. The outcome measures for this intervention were Activities specific balance confidence scale and berg balance scale.

ELIGIBILITY:
Inclusion Criteria:

* Elderly
* Both males and females were included in the study.
* Individuals with Mini Mental Status Examination score >23.
* History of falls in last 6 months

Exclusion Criteria:

* Any musculoskeletal disorder
* Any visual deficit
* Any systemic disease
* Any Neurological Disorder
* Any Cardiovascular and Respiratory Disorder
* Now cooperative Individuals
* Any Psychological disorder

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
BERG BALANCE SCALE | 6 weeks

SECONDARY OUTCOMES:
ACTIVITY BALANCE CONFIDENCE SCALE | 6 WEEKS

CONTACTS AND LOCATIONS:
Overall Officials: DIVYA MIDHA, MPT(NEURO), Principal Investigator — MAHARISHI MARKANDESHWAR UNIVERSITY

REFERENCES:
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568